CLINICAL TRIAL: NCT03611101
Title: Companion Protocol for the ¹³C-Methacetin Breath Test (MBT) for Use in Bristol-Myers Squibb Phase 2b Studies for BMS-986036 (PEG-FGF21), Under Studies Referenced in NCT03486899, NCT03486912
Brief Title: Companion Protocol for ¹³C-Methacetin Breath Tests in BMS: NCT03486899, NCT03486912 Referenced Trials
Status: Completed | Type: Interventional
Sponsor: Meridian Bioscience, Inc. (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: BMS-EX-0118
Record Dates: First submitted 2018-07-19; First posted 2018-08-02 (Actual); Results first posted 2022-08-09 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: NASH - Nonalcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Pegbelfermin

STUDY DESIGN:
Intervention Model Description: Subjects will be enrolled and randomized via interactive response technology (IRT) to receive BMS-9860936 Dose Level 1 , BMS-986036 Dose Level 2, BMS-9860936 Dose Level 3 or matching placebo in a 1:1:1:1 ratio. in both Stage 3 liver fibrosis and cirrhosis cohorts.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The collaborator is responsible for the masking process.
Oversight: Data Monitoring Committee: Yes | Unapproved Device: Yes

ARMS (4):
- BMS-986036 Dose Level 1 (Experimental): Administered by subcutaneous injection
  Interventions: Combination Product: ¹³C-Methacetin Breath Test; Drug: BMS-986036; Device: BreathID MCS device
- BMS-986036 Dose Level 2 (Experimental): Administered by subcutaneous injection
  Interventions: Combination Product: ¹³C-Methacetin Breath Test; Drug: BMS-986036; Device: BreathID MCS device
- BMS-986036 Dose Level 3 (Experimental): Administered by subcutaneous injection
  Interventions: Combination Product: ¹³C-Methacetin Breath Test; Drug: BMS-986036; Device: BreathID MCS device
- Placebo (Placebo Comparator): Administered by subcutaneous injection
  Interventions: Combination Product: ¹³C-Methacetin Breath Test; Drug: BMS-986036; Device: BreathID MCS device

INTERVENTIONS:
Combination Product: ¹³C-Methacetin Breath Test — A breath analyzer will be used to measure changes in 12C (carbon 12) to 13C (carbon 13) ratio as a result of metabolism of the Methacetin substrate before and after treatment.
Drug: BMS-986036 — Investigational drug for NASH treatment in Main BMS protocol
Device: BreathID MCS device — The BreathID MCS device is a breath analyzer specifically used for measuring changes in the ratio of 13CO2 and 12CO2 isotopes of carbon dioxide. The device is connected to the subject via a nasal cannula and breath is passively collected before and after ingestion of labelled 13C- Methacetin substrate.

SUMMARY:
This is a companion study assessing the ¹³C-Methacetin Breath Test (MBT) in subjects participating in the Bristol Myers-Squibb (BMS) NCT03486899 and NCT03486912 referenced studies using study drug BMS-986036.

DETAILED DESCRIPTION:
Subjects that are enrolled into either of two separate BMS sponsored IND (Investigational New Drug) studies (referenced by NCT03486899 and NCT03486912) at selected study sites will be offered the opportunity to perform the MBT. These will be considered as two separate study cohorts (cohort 1 and 2 respectively) within this companion protocol. There are four (4) treatment arms (BMS-986036 Dose Level 1, Dose Level 2, Dose Level 3 or matching placebo), as defined in the respective BMS sponsored protocols.

Cohort 1 consists of Subjects with NASH and stage 3 fibrosis, as assessed by a central laboratory reader of the liver biopsies (up to 160), and who meet all the NCT03486899 referenced study criteria.

Cohort 2 consists of Subjects with NASH and compensated liver cirrhosis, as assessed by a central laboratory reader of the liver biopsies (up to100), and who meet all the NCT03486912 referenced study criteria.

Approximately 75 sites will be included in the BMS studies, but not all participating sites will elect to perform the MBT. Each subject will perform up to 3 MBTs over 1 year; approximately one every 24 weeks.

The MBT in this study will only be conducted in the USA.

The primary purpose of the BMS study is to assess an experimental treatment for the following conditions: Hepatic cirrhosis, liver fibrosis, Nonalcoholic Fatty Liver Disease (NAFLD) and NASH (Nonalcoholic Steatohepatitis).

ELIGIBILITY:
Inclusion Criteria:

1. Liver biopsy performed within 6 months prior to the Screening Visit; if not performed within 6 months prior to the Screening Visit, a liver biopsy will be performed during the Screening Period and at least 4 weeks prior to randomization (Biopsy must be consistent with NASH, with: a) A score of at least 1 for each NAS component (steatosis, lobular inflammation, and ballooning), as assessed by the central reader AND b) Stage 3/Stage 4 (Cirrhosis) liver fibrosis (cohort 1 and cohort 2 respectively) according to the NASH CRN (Clinical Research Network) classification, as assessed by the central reader
2. Participants taking anti-diabetic, anti-obesity, or anti-dyslipidemic medications must have been on stable dosing regimens for at least 3 months prior to the Screening Visit
3. Participants taking vitamin E at doses ≥800 IU/day must have been on stable doses for at least 6 months prior to the Screening Visit (Vitamin E treatment must not have been initiated after the liver biopsy was performed)-

Exclusion Criteria:

1. Other causes of liver disease (e.g., alcoholic liver disease, hepatitis B virus infection, chronic hepatitis C virus infection, autoimmune hepatitis, drug-induced hepatotoxicity, Wilson disease, alpha-1-antitrypsin deficiency, iron overload, and hemochromatosis)
2. Current or past history of hepatocellular carcinoma (HCC)
3. Past or current evidence of hepatic decompensation (e.g., ascites, variceal bleeding, hepatic encephalopathy and/or spontaneous bacterial peritonitis) or liver transplantation Other protocol defined inclusion/exclusion criteria could apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2018-05-04 (Actual); Primary Completion 2020-08-18 (Actual); Study Completion 2021-11-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Spring Gastroenterology, Humble, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- BMS-986036 Dose Level 1 10 mg; BMS-986036 Dose Level 2 20 mg; BMS-986036 Dose Level 3 40 mg; Placebo: Administered by subcutaneous injection
  ¹³C-Methacetin Breath Test: A breath analyzer will be used to measure changes in 12C (carbon 12) to 13C (carbon 13) ratio as a result of metabolism of the Methacetin substrate before and after treatment.
  BMS-986036: Investigational drug for NASH treatment in Main BMS protocol
  BreathID MCS device: The BreathID MCS device is a breath analyzer specifically used for measuring changes in the ratio of 13CO2 and 12CO2 isotopes of carbon dioxide. The device is connected to the subject via a nasal cannula and breath is passively collected before and after ingestion of labelled 13C- Methacetin substrate.
Period: Overall Study
Arm/Group | BMS-986036 Dose Level 1 10 mg | BMS-986036 Dose Level 2 20 mg | BMS-986036 Dose Level 3 40 mg | Placebo
Started | 32 | 32 | 30 | 30
Completed | 25 | 28 | 27 | 23
Not Completed | 7 | 4 | 3 | 7

BASELINE CHARACTERISTICS:
Population: It should be noted, that there is no specific single outcome baseline measure, since the study compares each subject's baseline breath test results (PDR peak) to his/her future results to see if any changes were detected due to treatment. Every subject has a unique baseline. The actual measure is breath test PDR peak at Day 1. No analysis is done on the baseline measure , as it is only a reference for detecting changes.
Groups:
- Total: Total of all reporting groups
Arm/Group | BMS-986036 Dose Level 1 10 mg | BMS-986036 Dose Level 2 20 mg | BMS-986036 Dose Level 3 40 mg | Placebo | Total
Number analyzed (Participants) | 32 | 32 | 30 | 30 | 124
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.906 (6.981) | 58.438 (10.096) | 59.2 (9.034) | 60.433 (7.338) | 59.2 (8.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 20 | 17 | 17 | 78
  Male | 8 | 12 | 13 | 13 | 46
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 3 | 0 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 28 | 29 | 29 | 27 | 113
  More than one race | 4 | 0 | 1 | 3 | 8
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 32 | 32 | 30 | 30 | 124

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in MBT From Day 1 to Week 48
Description: Identification of subjects that experience a change in metabolic capacity in each of the treatment arms versus placebo arm after 48 weeks compared to baseline as determined independently by the Methacetin Breath Test (MBT) PDR peak output parameter under a responder analysis. No actual cut-off values or specific values of percent change criteria were pre-specified since this study was solely exploratory by nature as described in the protocol. The MBT PDR peak parameter was collected and analyzed for all those that performed the MBT based on the initial eligibility criteria of the study protocol and obtained a valid device printout with a PDR peak result, with no other methods or criteria used to exclude subjects. The outcome measure PDR peak is automatically calculated and generated in the printout when the device completes its measuring.
Time Frame: 48 weeks
Population: Percent Change in PDR peak (MBT parameter) from Day 1 to Week 48 in the Safety Analysis Set (Intended to be treated). Due to COVID-19, a follow up MBT at Week 48 was partial and did not include all those that performed the initial MBT on Day 1..
Measure: Mean (Standard Deviation); unit: percentage of change in MBT
Arm/Group | BMS-986036 Dose Level 1 10 mg | BMS-986036 Dose Level 2 20 mg | BMS-986036 Dose Level 3 40 mg | Placebo
Number analyzed (Participants) | 18 | 22 | 17 | 17
percentage of change in MBT | 8.8 (32.51) | 12.3 (33.36) | -4.7 (27.64) | 15.3 (31.58)

2. Secondary Outcome: Number of Subjects That Experience Deterioration Events
Description: Binary diagnosis of subjects that experience deterioration event as determined by the MBT compared to the placebo treatment arm
Time Frame: 48 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | BMS-986036 Dose Level 1 10 mg | BMS-986036 Dose Level 2 20 mg | BMS-986036 Dose Level 3 40 mg | Placebo
Number analyzed (Participants) | 32 | 32 | 30 | 30
Participants | 0 | 0 | 0 | 0

3. Secondary Outcome: Correlation
Description: Correlation of MBT PDR Peak to biopsy proven changes in fibrosis and/or NAS (NAFLD Activity Score) from Day 1 to Week 48. Total NAS score represents the sum of scores for steatosis (0-3), lobular inflammation (0-3), and ballooning (0-2), and ranges from 0-8; where 8 is the most severe.
Time Frame: 48 weeks
Measure: Number; unit: r-correlation
Groups:
- BMS-986036 Dose Level 1 10mg; BMS-986036 Dose Level 2 20 mg; BMS-968036 Dose Level 3 40 mg; Placebo: It should be noted that not all subjects had this NAS evaluation done and therefore there may be discrepancy between the amount of breath test performed and the the number of subjects with NAS evaluation.
Arm/Group | BMS-986036 Dose Level 1 10mg | BMS-986036 Dose Level 2 20 mg | BMS-968036 Dose Level 3 40 mg | Placebo
Number analyzed (Participants) | 9 | 12 | 8 | 10
r-correlation | -0.324 | -0.501 | 0.275 | -0.313

4. Secondary Outcome: Correlation
Description: Correlation of MBT changes to changes in liver stiffness as measured by Magnetic Resonance Elastography (MRE) from Day 1 to Week 48
Time Frame: 48 weeks
Measure: Number; unit: r-correlation
Groups:
- BMS-986036 Dose Level 1 10 mg; BMS-986036 Dose Level 2 20 mg; BMS-986036 Dose Level 3 40 mg; Placebo: It should be noted that not all subjects had this MRE evaluation done and therefore there may be discrepancy between the amount of breath test performed and the the number of subjects with MRE evaluation.
Arm/Group | BMS-986036 Dose Level 1 10 mg | BMS-986036 Dose Level 2 20 mg | BMS-986036 Dose Level 3 40 mg | Placebo
Number analyzed (Participants) | 13 | 15 | 13 | 16
r-correlation | 0.279 | -0.115 | -0.428 | 0.242

5. Secondary Outcome: Correlation
Description: Correlation of MBT changes to changes in Proton Density Fat Fraction (PDFF) as measured by Magnetic Resonance Imaging(MRI) from Day 1 to Week 48
Time Frame: 48 weeks
Measure: Number; unit: r-correlation
Groups:
- BMS-986036 Dose Level 1 10 mg; BMS-986036 Dose Level 2 20 mg; BMS-986036 Dose Level 3 40 mg; Placebo: It should be noted that not all subjects had this MRI evaluation done and therefore there may be discrepancy between the amount of breath test performed and the the number of subjects with MRI evaluation.
Arm/Group | BMS-986036 Dose Level 1 10 mg | BMS-986036 Dose Level 2 20 mg | BMS-986036 Dose Level 3 40 mg | Placebo
Number analyzed (Participants) | 16 | 21 | 14 | 17
r-correlation | -0.202 | -0.047 | 0.248 | -0.044

6. Secondary Outcome: Correlation
Description: Correlation of MBT changes to changes in Serum Pro-C3 results from Day 1 to Week 48
Time Frame: 48 weeks
Measure: Number; unit: r-correlation
Groups:
- BMS-986036 Dose Level 1 10 mg; BMS-986036 Dose Level 2 20 mg; BMS-986036 Dose Level 3 40 mg; Placebo: It should be noted that not all subjects had this Serum Pro-C3 evaluation done and therefore there may be discrepancy between the amount of breath test performed and the the number of subjects with Serum Pro-C3 evaluation.
Arm/Group | BMS-986036 Dose Level 1 10 mg | BMS-986036 Dose Level 2 20 mg | BMS-986036 Dose Level 3 40 mg | Placebo
Number analyzed (Participants) | 17 | 22 | 16 | 16
r-correlation | -0.001 | 0.242 | -0.263 | -0.072

7. Secondary Outcome: Correlation
Description: Correlation of MBT changes to changes in liver elastography by Fibroscan (in cohort 2 only) from Day 1 to Week 48
Time Frame: 48 weeks
Measure: Number; unit: r-correlation
Groups:
- BMS-986036 Dose Level 1 10 mg; BMS-986036 Dose Level 2 20 mg; BMS-986036 Dose Level 3 40 mg; Placebo: It should be noted that not all subjects had this Fibroscan evaluation done and therefore there may be discrepancy between the amount of breath test performed and the the number of subjects with Fibroscan evaluation.
Arm/Group | BMS-986036 Dose Level 1 10 mg | BMS-986036 Dose Level 2 20 mg | BMS-986036 Dose Level 3 40 mg | Placebo
Number analyzed (Participants) | 9 | 11 | 8 | 11
r-correlation | 0.491 | -0.351 | -0.121 | -0.43

8. Secondary Outcome: Correlation
Description: Correlation of MBT changes to changes in MELD (model for end-stage liver disease) scores (in cohort 2 only) from Day 1 to Week 48.The MELD score is generally calculated as: MELD = 3.78×ln[serum bilirubin (mg/dL)] + 11.2×ln[INR] + 9.57×ln[serum creatinine (mg/dL)] + 6.43. The higher the score, the more chances of mortality.
Time Frame: 48 weeks
Population: The objective of this endpoint was to compare changes in MBT collected for all subjects versus changes in MELD, a clinically used parameter used to assess liver function in each arm, over the course of the participation time in this trial, The result value is N/A if there were no subjects that had a MELD value that changed over the course of the trial, rendering r-correlation evaluation of changes in MBT versus changes in MELD not applicable.
Measure: Number; unit: r-correlation
Groups:
- BMS-986036 Dose Level 1 10 mg; BMS-986036 Dose Level 2 20 mg; BMS-986036 Dose Level 3 40 mg; Placebo: It should be noted that not all subjects had this MELD evaluation done and therefore there may be discrepancy between the amount of breath test performed and the the number of subjects with MELD evaluation.
Arm/Group | BMS-986036 Dose Level 1 10 mg | BMS-986036 Dose Level 2 20 mg | BMS-986036 Dose Level 3 40 mg | Placebo
Number analyzed (Participants) | 17 | 22 | 16 | 17
r-correlation | NA — The result value is N/A if there were no subjects that had a MELD value that changed over the course of the trial, rendering r-correlation evaluation of changes in MBT versus changes in MELD not applicable. | NA — The result value is N/A if there were no subjects that had a MELD value that changed over the course of the trial, rendering r-correlation evaluation of changes in MBT versus changes in MELD not applicable. | NA — The result value is N/A if there were no subjects that had a MELD value that changed over the course of the trial, rendering r-correlation evaluation of changes in MBT versus changes in MELD not applicable. | NA — The result value is N/A if there were no subjects that had a MELD value that changed over the course of the trial, rendering r-correlation evaluation of changes in MBT versus changes in MELD not applicable.

9. Secondary Outcome: Correlation
Description: Correlation of MBT changes to changes in CTP (Child-Turcotte-Pugh) score form Day 1 to Week 48. The CTP score is based on the sum of the ranges of the following parameters: total bilirubin (1-3), serum albumin (1-3), prothrombin time (1-3), ascites level (1-3) and hepatic encephalopathy grade (1-3). The higher the score, the more advanced is the liver disease
Time Frame: 48 weeks
Population: The objective of this endpoint was to compare changes in MBT collected for all subjects versus changes in CTP, a clinically used parameter used to assess liver function, in each arm, over the course of the participation time in this trial, The result value is N/A if there were no subjects that had a CTP value that changed over the course of the trial, rendering r-correlation evaluation of changes in MBT versus changes in CTP not applicable.
Measure: Number; unit: r-correlation
Groups:
- BMS-986036 Dose Level 1 10 mg: Level 1 10 mg Dose
- BMS-986036 Dose Level 2 20 mg: Dose Level 2 20 mg
- BMS-986036 Dose Level 3 40 mg: Dose Level 3 40 mg
- Placebo: Placebo
Arm/Group | BMS-986036 Dose Level 1 10 mg | BMS-986036 Dose Level 2 20 mg | BMS-986036 Dose Level 3 40 mg | Placebo
Number analyzed (Participants) | 32 | 30 | 30 | 30
r-correlation | NA — The result value is N/A if there were no subjects that had a CTP value that changed over the course of the trial, rendering r-correlation evaluation of changes in MBT versus changes in CTP not applicable. | NA — The result value is N/A if there were no subjects that had a CTP value that changed over the course of the trial, rendering r-correlation evaluation of changes in MBT versus changes in CTP not applicable. | NA — The result value is N/A if there were no subjects that had a CTP value that changed over the course of the trial, rendering r-correlation evaluation of changes in MBT versus changes in CTP not applicable. | NA — The result value is N/A if there were no subjects that had a CTP value that changed over the course of the trial, rendering r-correlation evaluation of changes in MBT versus changes in CTP not applicable.

ADVERSE EVENTS:
Time Frame: 48 hours after Methacetin Breath Test
Arm/Group | BMS-986036 Dose Level 1 10 mg | BMS-986036 Dose Level 2 20 mg | BMS-986036 Dose Level 3 40 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/32 | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/32 | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/32 | 0/32 | 0/30 | 0/30

LIMITATIONS AND CAVEATS:
This companion protocol, evaluating the utility of the MBT as a biomarker for assessment of treatment efficacy of the parent study drug, was designed to be exploratory by nature, and no pre-specified criteria for success were set a priori. The parent study conclusion was that the study drug is ineffective based on several standard clinically used biomarkers. As such, evaluating MBT as a biomarker of drug efficacy for a drug that was shown not to be effective is not applicable.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-02-20): https://cdn.clinicaltrials.gov/large-docs/01/NCT03611101/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-05): https://cdn.clinicaltrials.gov/large-docs/01/NCT03611101/SAP_001.pdf